CLINICAL TRIAL: NCT06005064
Title: The Effect of Krill Oil Supplementation on Muscle Function and Mass in Middle-aged Adults: A Randomised Controlled Trial
Brief Title: Middle Age muScle Krill Study
Acronym: MASK
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Glasgow (Other)
Responsible Party: Principal Investigator, Stuart Gray, Professor, University of Glasgow
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: MASK
Record Dates: First submitted 2023-08-16; First posted 2023-08-22 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Sarcopenia
Keywords: Krill oil; Muscle strength; Muscle mass; Middle-aged
MeSH Terms: conditions — Sarcopenia | interventions — Plant Oils

STUDY DESIGN:
Intervention Model Description: 1:1 basis
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Supplements will be identical in look and taste
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Krill oil 4g/day for 24 weeks
  Interventions: Dietary Supplement: Krill oil
- Placebo (Placebo Comparator): Vegetable oil 4g/day for 24 weeks
  Interventions: Dietary Supplement: Vegetable oil

INTERVENTIONS:
Dietary Supplement: Krill oil — Superba krill oil
  Arms: Intervention
Dietary Supplement: Vegetable oil — Mixed vegetable oil
  Arms: Placebo

SUMMARY:
This study will determine the effect of 6 months of supplementation with krill oil on muscle strength and mass in middle-aged adults. The study hypothesis is that krill oil supplementation will increase muscle strength and mass in middle-aged adults.

ELIGIBILITY:
Inclusion Criteria:

* Be 35-60 years old
* Have a BMI of less than 35kg/m2

Exclusion Criteria:

* People with diabetes, severe cardiovascular disease, seizure disorders, uncontrolled hypertension (>150/90mmHg at baseline measurement), cancer or cancer that has been in remission <5 years, ambulatory impairments which would limit the ability to perform assessments of muscle function, dementia, on anticoagulant therapy, and/or taking medication known to affect muscle (e.g., steroids).
* People who have allergies to seafood, and/or regular consumption of more than 1 portion of oily fish per week.
* People who perform regular (>1 day/week) resistance exercise training.

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 92 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Change in knee extensor maximal isometric torque ( MVC) | Change from baseline to 24 weeks
  Knee extensor maximal isometric torque measured during a maximal voluntary contraction

SECONDARY OUTCOMES:
Change in fat mass | Change from baseline to 24 weeks
  Whole body fat mass measured by measured via bio-electrical impedance
Change in lean mass | Change from baseline to 24 weeks
  Whole body lean mass measured by measured via bio-electrical impedance
Change in omega-3 levels | Change from baseline to 24 weeks
  Red blood cell omega-3 levels
Change in Grip strength | Change from baseline to 24 weeks
  Grip strength measured with a hand held dynamometer
Change in Muscle thickness | Change from baseline to 24 weeks
  Vastus lateralis muscle thickness measured by ultrasound

OTHER OUTCOMES:
Change in systemic inflammation | Change from baseline to 24 weeks
  Plasma levels of C-reactive protein, IL-1, IL-6, IL-8, IL-10, and TNF-α
Change in muscle inflammation | Change from baseline to 24 weeks
  Muscle total protein levels of TNF-α, IL-1β, IL-6, IL-8, MCP-1 and total and phosphorylated levels of NFκB, JNK1/2 and STAT3
Change in muscle anabolic signalling | Change from baseline to 24 weeks
  Muscle total and phosphorylated protein levels of mTOR, IRS-1, Akt, 4EBP-1, p70S6K, RPS6, FOXO-1, GSK3β and total protein levels of MAFBx and MURF-1

CONTACTS AND LOCATIONS:
Locations (1):
- University of Glasgow, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: No